CLINICAL TRIAL: NCT04319406
Title: Comparative Efficacy of Prolotherapy and Dry Needling in Management of Anterior Disc Displacement of Temporomandibular Joint
Brief Title: Comparative Efficacy of Prolotherapy and Dry Needling in Management of ADD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Jatin13
Record Dates: First submitted 2020-02-26; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Anterior Disk Displacement TMJ
MeSH Terms: interventions — Prolotherapy; Dry Needling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROLOTHERAPY (Experimental): Prolotherapy will be performed with 12.5 % Dextrose into superior joint space of involved TMJ
  Interventions: Procedure: Prolotherapy
- DRY NEEDLING (Active Comparator): Dry needling will be performed into superior joint space of involved TMJ
  Interventions: Procedure: Dry needling

INTERVENTIONS:
Procedure: Prolotherapy — Test group will be administered 12.5% Dextrose mainly into superior joint space according to symptoms of patient at baseline (0 week) and at biweekly intervals at 2 and 4 weeks i.e. a total of 3 injections. A 4th injection will be given at 6 weeks if required.
  Arms: PROLOTHERAPY
Procedure: Dry needling — Only dry needling will be performed at baseline (0 week) and at biweekly intervals at 2 and 4 weeks i.e. a total of 3 injections. A 4th injection will be given at 6 weeks if required.
  Arms: DRY NEEDLING

SUMMARY:
Pain and trismus caused by Anterior disc displacement ADD of temporomandibular joint (TMJ) are one of the prime concerns for the patients. In the recent times, Inflammatory Prolotherapy has been studied extensively and has produced promising results. In Inflammatory prolotherapy low grade inflammation is induced physiologically by injection of an irritant solution that initiates healing cascade which leads to repair of the joint structures.

Thus, the Present study is designed to evaluate the efficacy of dextrose prolotherapy for the treatment of ADD in TMJ.

DETAILED DESCRIPTION:
Temporomandibular joint (TMJ) is a ginglymodiarthroidal joint located bilaterally in the preauricular region of head. It is formed by the confluence of multiple skeletal, muscular, ligament and discal components which work in harmony with each other. Articular disc functions as a non-ossified bone, allowing complex movements, making it a compound joint.

Any loss in synchronization or harmony of the components of TMJ leads to temporomandibular disorders. Okeson broadly classified temporomandibular disorders into Masticatory muscle disorders, Temporomandibular joint disorders. Disc displacements are categorized under Temporomandibular joint disorders of the condyle-disc complex.

Normally articular disc is positioned over the cranial portion of mandibular condyle at 12 o'clock position when teeth are in occlusion. Abnormal position of disc with respect to mandibular condyle or mandibular fossa is known as disc displacement. Most common displacement of disc is in antero-medial direction.1 Disc displacements are of two types: disc displacement with reduction and disc displacement without reduction. Anterior disc displacement (ADD) associated with pain require treatment.

Established treatment modalities include use of Non steroidal anti inflammatory drugs (NSAIDS), Anterior repositioning appliances, Physiotherapy, Psychological therapy, Arthroscopy, Arthroplasty and Arthrocentesis. Newer treatment modalities that are under research are platelet rich plasma therapy, prolotherapy and stem cell therapy.

Prolotherapy, which is also known as regenerative injection therapy, and growth factor stimulation injection therapy. It can be used to strengthen and repair chronic ligament, joint, capsule, and tendinous injuries by stimulating proliferation of collagen at the fibro osseous junctions to promote soft tissue repair and relative pain.

Prolotherapy has recently emerged as a technique with low cost and minimal side effects for management of Temporomandibular joint disorders. Prolotherapy is of 3 types - Growth factor injection prolotherapy, growth factor stimulation prolotherapy and Inflammatory prolotherapy.2 In the recent times, Inflammatory Prolotherapy has been studied extensively and has produced promising results. In inflammatory prolotherapy low grade inflammation is induced physiologically by injection of an irritant solution that initiates healing process. Dextrose is most common and ideal proliferant used because it is a normal constituent of blood chemistry, water soluble and injected safely into multiple areas.3

The concentration of dextrose solution does not affect the results till the solution is hypertonic i.e above 10%. However, it is still not clear whether it is irritant effect of dextrose or mechanical injury caused by needle that produce the desired result .2 Dry needling can also induce a low grade inflammatory process in the joint. Dry needling has been proven to be equally beneficial in temporomandibular myofascial pain that involves inserting a needle into trigger points to inactivate them. Stimulation of these trigger points by needling alone, produce an analgesic effect by altering somatosensory thresholds .4 So, the present study has been designed to compare the efficacy of dextrose solution injection compared to dry needling in ADD of TMJ.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with Anterior disc displacement clinically according to TMD/RDC criteria (2013-14).
2. Patients diagnosed with Anterior disc displacement confirmed using Magnetic Resonance Imaging.

Exclusion Criteria:

1. Patients with phobia to needles
2. Patients who have undergone previous treatment for anterior disc displacement in past 6 months
3. Patients who are allergic to the components of prolotherapy solution
4. Patients with active infection at the site of injection
5. Patients on anticoagulant medication
6. Patients with healing disorder or systemic disease where healing response is compromised
7. Patients with epilepsy/seizures
8. Patients with bleeding and clotting disorder
9. Patients with malignancy
10. Patients with uncontrolled para-functional habits

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-05 (Actual); Primary Completion 2020-08-05 (Estimated); Study Completion 2020-09-05 (Estimated)

PRIMARY OUTCOMES:
Intensity of pain | 6 months
  VAS Score
Maximal mouth opening | 6 months
  Manual measurement in mm

SECONDARY OUTCOMES:
Range of Right and left Lateral excursion movements | 6 months
  Manual measurement in mm
Range of Protrusive movement | 6 months
  Manual measurement in mm
Joint sounds | 6 months
  Presence or absent
Pain medicine utilization | 6 months
  No. of tablets consumed
Patient satisfaction | 6 months
  Likert scale
Assessment of Sleep pattern | 6 months
  VAS score

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India